CLINICAL TRIAL: NCT06404086
Title: RECOVER-SLEEP: A Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-SLEEP: Platform Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112484; OTA-21-015G (Other Grant/Funding Number: NIH Grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-06; First posted 2024-05-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Long COVID; Long COVID-19; Hypersomnia; Sleep Disturbance
Keywords: PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Disorders of Excessive Somnolence; Parasomnias | interventions — Modafinil; solriamfetol; Melatonin

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an intervention appendix based on their symptoms of sleep disturbance. Within the appendix, participants will be randomly assigned based on the appendix study design. Site investigators and personnel will be informed as to which study intervention appendix participants are assigned, but they will be blinded to whether participants are receiving the active study intervention or control, when possible. Similarly, participants will be blinded to active intervention or control, when possible. Randomization will be stratified by the study site; other stratification factors may be considered per appendix.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hypersomnia Arm (Appendix A) (Other): This is a double-blind, phase 2, randomized, placebo-controlled interventional trial of a wake-promoting drug (modafinil or solriamfetol) to treat hypersomnia, defined by elevated scores (> 55) on the PROMIS 8a SRI scale, in participants with PASC. Participants will be randomized to study drug or control. Participants who meet the eligibility criteria for modafinil will receive either active modafinil or modafinil-matched control. If modafinil is contraindicated, participants will be assessed for solriamfetol. If participants are eligible for solriamfetol, they will receive either active solriamfetol or solriamfetol-matched control. If solriamfetol is contraindicated, participants will be excluded from Appendix A. Modafinil and solriamfetol will be analyzed as a single wake-promoting drug condition versus control. The intervention duration will be 10 weeks.
  Anticipated enrollment is 474 participants. Details about the Hypersomnia Appendix are available under NCT06404099.
  Interventions: Drug: Modafinil; Drug: Modafinil Placebo; Drug: Solriamfetol; Drug: Solriamfetol Placebo
- Complex PASC related Sleep Disturbances (CPSD) Arm (Appendix B ) (Other): This is a double-blind, phase 2, randomized, placebo-controlled, interventional trial that combines brief education and a tailored sleep timing prescription for CPSD with therapies that modify circadian timing for participants who report poor sleep quality or daytime sleep-related impairment, defined by elevated scores (≥55) on the PROMIS 8b SD scale, in participants with symptoms that occurred or worsened after COVID-19 infection. Interventions involve tailored lighting (TL) and melatonin. Participants will be randomly assigned to 1 of 4 groups: (a) active TL + oral melatonin, (b) active TL + placebo melatonin, (c) placebo TL + oral melatonin, and (d) placebo TL + placebo melatonin. All groups will receive BBT-CPSD. It is a 2x2 factorial design schema. The intervention duration will be 8 weeks.
  Anticipated enrollment for this appendix is 600 participants. Additional details about the CPSD Appendix are available under NCT06404112.
  Interventions: Drug: Melatonin; Drug: Melantonin Placebo; Device: Tailored lighting (TL) Active; Device: Tailored lighting (TL) Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil is used off-label based on supporting published evidence in major depressive disorder (antidepressant augmentation), multiple sclerosis-related fatigue, Parkinson disease-related excessive daytime sleepiness, and severe cancer-related fatigue (in patients receiving active treatment). Doses up to 400 mg/day, given as a singleMode dose, have been well tolerated, but there is no consistent evidence that this dose confers additional benefit beyond that of the 200 mg dose.
  Study drug administration will total 10 weeks.
  Arms: Hypersomnia Arm (Appendix A)
Drug: Modafinil Placebo — The placebo will be tooled to look similar to the modafinil tablet, but it will not contain the active ingredient. Modafinil placebo dosing will follow the same titration scheme as modafinil treatment.
  Unblinded study personnel will manage modafinil and placebo disbursement to maintain blinding among participants and blinded study personnel, including site investigators.
  Arms: Hypersomnia Arm (Appendix A)
Drug: Solriamfetol — The proposed doses and the schedule of dose escalation are consistent with currently approved FDA labeling for solriamfetol for other disorders of excessive daytime sleepiness.
  Solriamfetol dosing will total 10 weeks, including 3 weeks for titration and 7 weeks of maintenance. Solriamfetol will be given as a 75 mg tablet (1 or 2 per day) in the morning. The 3-week titration will be facilitated by phone calls between the study team and participants. Titrations in dose will be dependent upon participants' symptoms and tolerance to solriamfetol, with a goal of participants taking the highest dose permitted by symptoms. This dose will be used for the maintenance phase.
  Arms: Hypersomnia Arm (Appendix A)
Drug: Solriamfetol Placebo — The placebo tablet will be tooled to look similar to the solriamfetol tablet, but it will not contain the active ingredient. Solriamfetol placebo dosing will follow the solriamfetol dosing scheme and goal.
  Unblinded study personnel will manage solriamfetol and placebo disbursement to maintain blinding among participants and blinded study personnel, including site investigators.
  Arms: Hypersomnia Arm (Appendix A)
Drug: Melatonin — Melatonin dosing will be one tablet of 3 mg immediate release daily consumed 2 hours before the participant's desired bedtime, which is defined as the time at which the participant tries to fall asleep.
  Arms: Complex PASC related Sleep Disturbances (CPSD) Arm (Appendix B )
Drug: Melantonin Placebo — Melatonin placebo dosing will be one placebo tablet once daily consumed 2 hours before the participant's desired bedtime.
  Arms: Complex PASC related Sleep Disturbances (CPSD) Arm (Appendix B )
Device: Tailored lighting (TL) Active — TL will be delivered similarly to both active and placebo groups, but the circadian stimulus (the amount of light) will be different, albeit practically unidentifiable to participants.
  Arms: Complex PASC related Sleep Disturbances (CPSD) Arm (Appendix B )
Device: Tailored lighting (TL) Placebo — TL will be delivered similarly to both active and placebo groups, but the circadian stimulus (the amount of light) will be different, albeit practically unidentifiable to participants.
  Arms: Complex PASC related Sleep Disturbances (CPSD) Arm (Appendix B )

SUMMARY:
The platform protocol is designed to be flexible so that it is suitable for a range of study settings and intervention types. Therefore, the platform protocol provides a general protocol structure that can be shared by multiple interventions and allows comparative analysis across the interventions. For example, objectives, measures, and endpoints are generalized in the platform protocol, but intervention-specific features are detailed in separate appendices.

This platform protocol is a prospective, multi-center, multi-arm, randomized controlled platform trial evaluating potential interventions for PASC-mediated sleep disturbances. The hypothesis is that symptoms of sleep and circadian disorders that emerge in patients with PASC can be improved by phenotype-targeted interventions. Specific sleep and circadian disorders addressed in this protocol include sleep-related daytime impairment (referred to as hypersomnia) and complex PASC-related sleep disturbance (reflecting symptoms of insomnia and sleep-wake rhythm disturbance).

DETAILED DESCRIPTION:
Interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix.

After completing Baseline assessments, participants will be randomized to an intervention group, which is based on their sleep phenotype, or into a placebo/control group.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. ≥ 18 years of age at the time of enrollment
2. Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization:

   Suspected* case of SARS-CoV-2 infection - Three options, A through C:

   A. Met the clinical OR epidemiological criteria:
   1. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia;
   2. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or B. Presented with acute respiratory infection with a history of fever or measured fever of ≥ 38°C and cough, with onset within the last 10 days, and required hospitalization; or C. Presented with no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.

   Probable* case of SARS-CoV-2 infection, defined as having met the clinical criteria above AND was a contact of a probable or confirmed case or is linked to a COVID-19 cluster; or

   Confirmed case of SARS-CoV-2 infection - Two options, A through B:

   A. Presented with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or B. Met clinical criteria AND/OR epidemiological criteria (See suspected case A), with a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.

   * Suspected and probable cases will only be allowed if they occurred before May 1, 2021, and will be limited to 10% of the study population. Otherwise, confirmed cases are required.
3. New/worse sleep problems following a SARS-CoV-2 infection that have persisted for at least 12 weeks and are still present at the time of consent
4. PROMIS 8a SRI or 8b SD T Score ≥ 55**

   ** Screening with both the PROMIS 8a SRI and 8b SD will occur for the phenotype assessment portion of the protocol.
5. Willing and able to provide informed consent, complete the surveys and clinical assessments, and return for all of the necessary follow-up visits
6. Adequate method of birth control for participants of child-bearing potential

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known active acute SARS-CoV-2 infection ≤ 4 weeks from consent
2. Known pregnancy, breastfeeding, or contemplating pregnancy during the study period
3. Untreated sleep apnea (AHI ≥ 15 or severe sleep-related hypoxemia)
4. Current night or rotating shift work
5. Known history of narcolepsy prior to SARS-CoV-2 infection
6. Any non-marijuana illicit drug use within 30 days of informed consent
7. Known history of severe mental disorder, such as psychotic disorders and bipolar disorder
8. Current or recent use (within the last 14 days) of study intervention or similar intervention to treat the underlying condition, unless a washout period is permitted per appendix*
9. Known allergy/sensitivity or any hypersensitivity to components of the study intervention or control*
10. Known contraindication(s) to study intervention including prohibited concomitant medications and without the ability to safely hold prohibited concomitant medications (see appendices)*
11. Currently receiving/using intervention from another clinical trial that could impact or mask treatment effect; refer to MOP for details
12. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

(*)If only one study intervention appendix is open at the time of enrollment. If multiple study intervention appendices are open, a participant may be excluded from any study intervention appendix based on contraindications listed in the study intervention appendix, current use of study intervention, or known allergy/sensitivity/hypersensitivity yet remain eligible for the remaining study intervention appendices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of participants enrolled in each Appendix | 12 months
  Total number of participants enrolled in each Appendix will be reported. Appendix-specific outcome measure data will be reported under the associated NCT#.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Barkauskas, MD, Study Chair — Duke Clinical Research Institute; Susan Redline, MD MPH, Study Chair — Brigham and Women's Hospital
Locations (47):
- United States (47):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona Banner Medical Center, Tucson, Arizona
  - The Southern Arizona VA Health Care System, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - University of California San Francisco General Hospital, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Hope Clinic, Decatur, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Cook County Health Specialty Care Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Rutgers University - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Southwest Family Medicine Associates, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - New Dawn Wellness and Medical Research Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - University Physicians and Surgeons (DBA Marshall Health), Huntington, West Virginia
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
The summary of results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT06404086/ICF_000.pdf